CLINICAL TRIAL: NCT01070654
Title: Prospective, Open, Uncontrolled, Non-randomized and Monocentric Trial on the Efficacy and the Inflammatory Effects of a Lung Recruitment Manoeuvre in Mechanical Ventilated Patients With Respiratory Failure
Brief Title: Inflammatory Effects of a Lung Recruitment Manoeuvre
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Dr Francesco Forfori, UO IV Anestesia e Rianimazione
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM0910; RMSGMFF (Other: IV Anestesia e Rianimazione)
Record Dates: First submitted 2010-02-16; First posted 2010-02-18 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-02

CONDITIONS: Respiratory Insufficiency; Respiratory Distress Syndrome, Adult
Keywords: ARDS; Recruitment Manoeuvres; PEEP; Cytokines; Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 40/30 Recruitment Manoeuvre (Experimental): Patients with respiratory failure that will be first ventilated for 30 minutes according to standardized baseline protective ventilation and after that will receive the recruitment manoeuvre
  Interventions: Procedure: 40/30 recruitment manoeuvre; Device: continuous positive airway pressure (CPAP)

INTERVENTIONS:
Procedure: 40/30 recruitment manoeuvre — The ventilator will be switched to the continuous positive airway pressure (CPAP) mode and the pressure will be increased to 40 cmH20 for 30 seconds.
  Other Names: Recruitment Manoeuvres; ARDS open lung strategy; PEEP
Device: continuous positive airway pressure (CPAP) — continuous positive airway pressure (CPAP)

SUMMARY:
Recruitment manoeuvres, consisting of sustained inflations at high airway pressures, have been advocated as an adjunct to mechanical ventilation in lung protective ventilation strategies to prevent the collapse of the lung.

This study aims to determine the safety and efficacy of a recruitment manoeuvre, by considering its impact on gas exchange, hemodynamics and on the release of systemic inflammatory mediators.

DETAILED DESCRIPTION:
This prospective study will analyse the effects of a single recruitment manoeuvre in critically ill patients. Subjects will be mechanically ventilated patients needing alveolar RMs. After a period of stable lung protective approach ventilation, they will receive the "40/30" RM; lung mechanics, gas exchange, hemodynamics and plasmatic concentration of inflammatory mediators will be obtained before and after the RM. An ultrasound score, established from the lung aeration status of upper and lower parts of anterior and lateral chest wall, will also be calculated before and after the manoeuvre.In selected patients cytokine release in the bronchoalveolar lavage will be measured as well.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical Ventilation
* Arterial catheter inserted
* Hypoxemic respiratory failure (Pa02/FiO2 <300)
* Radiological evidence of atelectasis or pulmonary infiltrates in the CXR
* Informed consent

Exclusion Criteria:

* Elevated intracranial pressure >25 mmHg
* Bronchopulmonary fistula
* Emphysema
* Kidney or Liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Plasmatic concentration of inflammatory mediators IL-1, IL-6, IL-8, IL-10, TNFa | T0 (baseline), T4 (3 hrs), T5 (12 hrs)
Plasmatic concentration of Nitric Oxide | T0 (baseline), T6 (24 hrs)
Lung mechanics (Peak pressure, Mean pressure, Compliance, Resistance) Gas exchange (pH, PaO2, PaCO2, HCO3-, SaO2, PaO2/FiO2) Haemodynamics (Mean arterial pressure, Heart rate) | T0 (baseline), T1 (30 secs), T2 (1 hr), T3 (2 hrs)
Echographic score of lung aeration | T0 (baseline), T2 (1 hr), T4 (3 hrs)
Chest X-Ray | T6 (24 hrs)

SECONDARY OUTCOMES:
Levels of IL-1, IL6, IL-8, IL-19, TNFa in the bronchoalveolar lavage | T0 (baseline), T4 (3 hrs)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Forfori, Principal Investigator — UO IV Anestesia e Rianimazione
Locations (1):
- U.O. Anestesia e Rianimazione IV, Azienda Ospedaliero Universitaria Pisana, Pisa, Pisa, Italy